CLINICAL TRIAL: NCT02808195
Title: Comparative Effectiveness of a Kinect-based Unilateral Arm Training System vs Constraint-Induced Therapy for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201601057RINB
Record Dates: First submitted 2016-05-24; First posted 2016-06-21 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Neurological Rehabilitation; Upper Extremity
MeSH Terms: conditions — Cerebral Palsy | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- constraint-induced therapy (Experimental): training of the more affected arm and restraint the less affected arm
  Interventions: Other: Constraint-induced therapy
- kinect-based constraint-induced therapy (Experimental): training of the more affected arm and restraint the less affected arm by kinect-game
  Interventions: Other: kinect-based constraint-induced therapy

INTERVENTIONS:
Other: Constraint-induced therapy
  Arms: constraint-induced therapy
Other: kinect-based constraint-induced therapy
  Arms: kinect-based constraint-induced therapy

SUMMARY:
The aims of the present study is to evaluate the effectiveness of Kinect-based upper limb motor rehabilitation system (ULMTS) program on motor performance and functional outcomes.

DETAILED DESCRIPTION:
The specific aims of this study project will be:

To compare the effectiveness of intervention groups using Kinect-based ULMTS with constraint-induced therapy on motor improvement in children with hemiplegic CP. The investigators hypothesize that motor improvement in using Kinect-based ULMTS will be comparable to constraint-induced therapy.

ELIGIBILITY:
Inclusion criteria are:

1. 3-16 years old
2. diagnosed with congenital hemiplegic or CP with one more affected side
3. considerable nonuse of the affected upper limb.

Exclusion criteria are:

1. no excessive muscle tone (Modified Ashworth Scale ≤ 2 at any joints of the upper limb) before beginning treatment (Bohannon & Smith, 1987)
2. no severe cognitive, visual, or auditory disorders according to medical documents, parental reports, and the examiner's clinical observation
3. no injections of botulinum toxin type A or operations on the upper limb within 6 months.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Performance Change assessed by Kinematic analysis | baseline, 2 months and 6 months
  Kinematic analysis including measuring the parameters of endpoint control, joint recruitment and inter-joint coordination, and trunk involvement.

SECONDARY OUTCOMES:
score change of Bruininks-Oseretsky Test of Motor Proficiency Second Edition (BOT-2) | baseline, 1 months, 2 months and 6 months
score change of Melbourne Assessment 2 (MA2) | baseline, 1 months, 2 months and 6 months
score change of Pediatric Motor Activity Log-Revised (PMAL-R) | baseline, 1 months, 2 months and 6 months
score change of ABILHAND-kids | baseline, 1 months, 2 months and 6 months
score change of Functional Independence Measures for children (WeeFIM) | baseline, 1 months, 2 months and 6 months
score change of Pediatric evaluation of disability inventory (PEDI) | baseline, 1 months, 2 months and 6 months
score change of Cerebral Palsy Quality of Life Questionnaire for Children (CP-QOL) | baseline, 1 months, 2 months and 6 months
score change of Test of Visual Perceptual Skills-3rd (TVPS-3) | baseline, 1 months, 2 months and 6 months
score change of Test of Playfulness (TOP) | baseline, 1 months, 2 months and 6 months
score change of Engagement Questionnaire (EQ) | baseline, 1 months, 2 months and 6 months
score change of Clint Satisfaction Questionnaire (CSQ) | baseline, 1 months, 2 months and 6 months
score change of Parenting Stress Index-Short Form (PSI-SF) | baseline, 1 months, 2 months and 6 months
Muscle strength | baseline, 2 months and 6 months
  measured by electromyography
score change of Building Tower Test | baseline, 1 months, 2 months and 6 months
score change of Test of String Beads | baseline, 1 months, 2 months and 6 months
score change of Box and Block Test | baseline, 1 months, 2 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Ling Chen, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Shih TY, Wang TN, Shieh JY, Lin SY, Ruan SJ, Tang HH, Chen HL. Comparative effects of kinect-based versus therapist-based constraint-induced movement therapy on motor control and daily motor function in children with unilateral cerebral palsy: a randomized control trial. J Neuroeng Rehabil. 2023 Jan 27;20(1):13. doi: 10.1186/s12984-023-01135-6. PMID 36703170
- [Derived] Chen HL, Lin SY, Yeh CF, Chen RY, Tang HH, Ruan SJ, Wang TN. Development and Feasibility of a Kinect-Based Constraint-Induced Therapy Program in the Home Setting for Children With Unilateral Cerebral Palsy. Front Bioeng Biotechnol. 2021 Oct 26;9:755506. doi: 10.3389/fbioe.2021.755506. eCollection 2021. PMID 34765593